CLINICAL TRIAL: NCT06451640
Title: A Multicenter, Randomized, Ongoing Trial Evaluating the Long-term Safety and Efficacy of TQC2731 Injection in the Treatment of Chronic Sinusitis With Nasal Polyps
Brief Title: A Extension Clinical Study of TQC2731 Injection in the Treatment of Chronic Sinusitis With Nasal Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-II-03
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 210mg of TQC2731 injection (Experimental): 210mg of TQC2731 injection combined with Mometasone Furoate Aqueous Nasal Spray, 28days as a treatment cycle.
  Interventions: Drug: 210mg of TQC2731 injection
- 420mg of TQC2731 injection (Experimental): 420mg of TQC2731 injection combined with Mometasone Furoate Aqueous Nasal Spray, 28days as a treatment cycle.
  Interventions: Drug: 420mg of TQC2731 injection

INTERVENTIONS:
Drug: 210mg of TQC2731 injection — TQC2731 injection is a thymic stromal lymphopoietin (TSLP) monoclonal antibody.
  Arms: 210mg of TQC2731 injection
Drug: 420mg of TQC2731 injection — TQC2731 injection is a thymic stromal lymphopoietin (TSLP) monoclonal antibody.
  Arms: 420mg of TQC2731 injection

SUMMARY:
This study aims to evaluate the efficacy and safety of TQC2731 injection in the treatment of chronic sinusitis with nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign informed consent before study, fully understand the purpose, procedures and possible adverse reactions of the study;
* Male and female, ≥18 years old;
* Participate in the clinical study of TQC2731 for the treatment of chronic rhinosinusitis with nasal polyps (CRSwNP) (study number TQC2731-II-02) and meet the following criteria "a" or "b": a. Participants complete the prescribed treatment according to the protocol requirements and complete end of treatment (EOT) visits; b. The subject withdrew early due to poor compliance or other objective reasons other than TQC2731 related adverse events (AEs), and completed the early withdrawal visit according to the plan. After evaluation by the researcher and sponsor, the factors that led to the subject's early termination of the main study treatment have disappeared/no longer affect the subject's participation in this continuing study;
* Subjects used steady dose of intranasal glucocorticoids (INCS) over 4 weeks before screening (subjects willing to use Mometasone Furoate Aqueous Nasal Spray (MFNS) while studying);
* Subjects agree from sign informed consent to last administration over 6 mouth without Family planning，and take effective non-pharmaceutical contraception.

Exclusion Criteria:

* In the main study (TQC2731-II-02), SAE related to TQC2731 occurred, or TQC2731 treatment was terminated due to AE related to TQC2731. After discussion between the investigator and the sponsor, it was determined that the subject was not suitable to continue receiving TQC2731 treatment;
* The subjects had poor compliance in the main study and were deemed unable to complete this continuing study by the researchers;
* During the main study (TQC2731-II-02), any serious progression or poorly controlled comorbidities were found (such as asthma exacerbation requiring adjustment of background medication), and the main investigator determined that the subject was not suitable to participate in the trial;
* Presence of conditions/concomitant diseases that affect the evaluation of efficacy, e.g.

  1. Posterior nostril polyps;
  2. Imaging suspected or confirmed fungal sinusitis;
  3. Nasal polyp score(NPS) cannot be evaluated due to nasal surgery to alter the structure of the lateral nasal wall;
  4. Subjects with nasal malignancies and benign tumors (papilloma, blood furuncle, etc.).
* Any type of active malignancy or a history of malignancy (Patient with basal cell carcinoma, skin localized squamous cell carcinoma or carcinoma in situ of cervix, if curative treatment was completed for more than 12 months prior to visit 1 can join the study; Other malignant tumors can join the study if patients had completed curative therapy for at least 5 years prior to visit 1);
* Active autoimmune disease;
* Known or suspected history of immunosuppression, immune dysfunction, or immune dysfunction, including but not limited to invasive opportunistic infections, even if the infection has subsided;
* Uncontrolled epistaxis occurred within 2 months before screening;
* Infection requiring treatment with systemic antibacterial, antiviral, antifungal, antiparasitic, or antiparasitic agents occurred within 14 days before screening;
* Helminth parasite infection was diagnosed within 24 weeks prior to screening and had not received or failed to respond to standard treatment;
* Leukotriene antagonists/modulators were used while screening(using a stable dose of leukotriene modulator for ≥30 days before screening was accepted);
* Regular use of decongestants (topical or systemic) before screening, short-term use for endoscopy excepted;
* Patients who received any of the following treatments before screening:

  1. Immunosuppressive therapy had been administered within the previous 8 weeks or five half-lives (whichever was longer), (including but not limited to cyclophosphamide, cyclosporine, interferon-γ, azathioprine, methotrexate, mycophenolate mofetil and tacrolimus, etc.);
  2. Monoclonal antibody therapy had been administered within the previous 8 weeks or five half-lives (whichever was longer), (Including but not limited to: benralizumab, mepolizumab, omalizumab, resveratrol, dupilumab, etc.);
  3. Systemic glucocorticoids were used during the first 28 days;
  4. Glucocorticoid-eluting nasal stents were used during the first 6 mouths;
  5. Immune globulin or blood products therapy were used during the first 28 days; 6）Live attenuated vaccine was administered for the first 28 days or during the planned study period; 7）Received allergen specific immunotherapy 6 mouth before screening(if being treated at a stable dose and not expected to change during study,3 mouth before screening and 1 mouth before visit 1 were accepted); 8）Join any other study within 3 mouths.
* Patients with concomitant asthma begin inhaled corticosteroid therapy within the first 4 weeks of the screening period (For patients who have been assessed to maintain a stable dose for at least 4 weeks prior to screening and whose dose has been maintained throughout the entire study period, inhaled corticosteroids can be administered at a dose of ≤ 1000μ Fluticasone propionate or equivalent doses of other inhaled corticosteroids.);
* Any infectious disease screening indicator that meets the following criteria during screening:

  1. Active tuberculosis infection during screening;
  2. Hepatitis B virus surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and hepatitis B virus (HBV) DNA positive;
  3. Anti-hepatitis C virus (Anti-HCV) positive and Hepatitis C virus ribonucleic acid (HCV-RNA) positive;
  4. Positive Treponema pallidum antibody (Anti TP) (if the Treponema pallidum serological test is positive, further non treponema pallidum serological tests will be conducted, the latter being negative and judged by the researcher as a patient who has previously been infected with syphilis but has been cured and meets the inclusion criteria);
  5. Positive for human immunodeficiency virus antibodies (Anti HIV);
* Abnormal laboratory test results:

  1. Aspartate aminotransferase (AST)>2.5 x upper limit of normal value (ULN);
  2. Alanine aminotransferase (ALT)>2.5 x upper limit of normal value (ULN);
  3. Creatinine>1.5 x ULN.
* Pregnant or lactating women;
* A history of or allergic reaction to Mometasone furoate nasal spray (Nasonex ®) or any component of TQC2731 injection;
* A history of systemic allergy to any biologic drug(except local injection site reactions);
* The subjects had poor compliance and were judged unable to complete the study;
* Any clinically significant abnormal findings, including physical examination, vital signs, 12-lead electrocardiogram, blood biochemistry, blood routine or urine routine, and the researcher's judgment that participating in the trial may put the patient at risk, or may affect the study results or hinder the patient's ability to complete the entire study process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse event rate | Up to thirty six weeks
  The frequency of treatment-related adverse events (TEAEs) occurring during treatment at each evaluation time point.

SECONDARY OUTCOMES:
Treatment-related serious adverse events rate | Up to thirty six weeks
  The frequency of serious adverse events (SAEs) occurring during treatment at each evaluation time point.
Abnormal laboratory test indicators | Up to thirty six weeks
  The number and severity of abnormal laboratory test indicators.
Nasal Polyp Score (NPS) | Baseline up to thirty six weeks
  NPS is the sum of the left and right nostril scores evaluated through nasal endoscopy, with a total score range of 0 to 8. NPS is based on polyp grading, with a score of 0-4 based on polyp grading.
Nasal congestion score (NCS) | Baseline up to thirty six weeks
  NCS is determined by the subjects based on the severity of the nasal congestion in the past 24 hours. This score uses a 0-3 classification scale, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, and 3=severe symptoms.
Anosmia score | Baseline up to thirty six weeks
  Anosmia Score is evaluated by subjects based on their severity of Anosmia on the day. This score uses a 0-3 classification scale, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, and 3=severe symptoms.
Total symptom score (TSS) | Baseline up to thirty six weeks
  TSS is the sum of nasal congestion, anosmia, and rhinorrhea (the average of anterior and posterior rhinorrhea), with a score range of 0-9 points. The severity is evaluated by the subject and recorded on the subject diary record card.
Visual analogue scale (VAS) for sinusitis | Baseline up to thirty six weeks
  VAS for sinusitis is a questionnaire that subjective evaluation of the overall severity of sinusitis by subjects, with a score range of 0-10 points. The higher the score, the greater the impact of sinusitis on the quality of life of the subjects.
Lund Mackay (LMK) score | Baseline up to twenty eight weeks
  The LMK score is based on the results of sinus Computed Tomography (CT) scans. Evaluated by researchers, divided into left and right sinus systems, with 0-12 points per side and a total score of 0-24 points.
Immunogenicity-anti-drug antibody | 1 hour on day 1 before administration, day 197, day 253 during withdrawal
  Incidence and their titers of Anti-drug antibody (ADA).
Immunogenicity-neutralizing antibody | 1 hour on day 1 before administration, day 197, day 253 during withdrawal
  Incidence of neutralizing antibody (Nab).

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital Of Dalian university, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - The Afiliated Hospital Of QINGDAO University, Qingdao, Shandong
  - Eye＆Ent Hospital of Fudan University, Shanghai, Shanghai Municipality
  - ChengDu Second People's Hospital, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang